CLINICAL TRIAL: NCT02045394
Title: Multicenter, Prospective, Observational Study on Epidemiology and Diagnosis of Haemoptysis
Brief Title: Epidemiology and Diagnosis of Haemoptysis: a Multicenter Study
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Fabiano Di Marco, M.D., Ph.D., University of Milan
Other Study IDs: HAEMOPTYSIS76
Record Dates: First submitted 2014-01-13; First posted 2014-01-24 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Lung Cancer; Tuberculosis; Bronchiectasis; Pneumonia; Acute Bronchitis; Chronic Obstructive Pulmonary Disease; Cryptogenic Haemoptysis
Keywords: haemoptysis; hemoptysis; airway bleeding
MeSH Terms: conditions — Lung Neoplasms; Tuberculosis; Bronchiectasis; Pneumonia; Bronchitis; Pulmonary Disease, Chronic Obstructive; Hemoptysis | interventions — X-Rays; Bronchoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients presenting with haemoptysis
  Interventions: Other: Chest X-ray; Other: computed tomography of the chest; Procedure: Bronchoscopy

INTERVENTIONS:
Other: Chest X-ray
Other: computed tomography of the chest
  Other Names: chest CT scan
Procedure: Bronchoscopy — In patients with haemoptysis bronchoscopy will be performed with flexible bronchoscope. A systemic research of bleeding site and causes will be done. Microbiological or pathological sampling will be executed if clinically required. In selected patients, bronchoscopy might be performed with the rigid instrument or the flexible bronchoscope in intubated patients.

SUMMARY:
Haemoptysis is the coughing up of blood originating from the respiratory tract. It is a common and worrying clinical symptom which can be due to different aetiologies including lung cancer, tuberculosis, COPD, bronchiectasis, pneumonia, acute bronchitis or unknown origin (cryptogenic haemoptysis). Epidemiology and optimal diagnostic approach are largely unclear. Aims of this study are to define current epidemiology and to provide the best diagnostic approach by providing a diagnostic algorithm.

ELIGIBILITY:
Inclusion Criteria:

* haemoptysis requiring a diagnosis

Exclusion Criteria:

* history of known bleeding lesions in the upper or lower airways

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients and outpatients with haemoptysis requiring a diagnosis referred for medical consultation to italian university and clinical hospitals.
Sampling Method: Probability Sample
Enrollment: 610 (Actual)
Dates: Start 2013-06; Primary Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Percentage of patients presenting with haemoptysis affected by lung cancer, tuberculosis, bronchiectasis, pneumonia, acute bronchitis, cryptogenic haemoptysis or other causes. | 18 months
  To define the prevalence of diseases presenting with haemoptysis by measuring percentage of patients presenting with haemoptysis affected by lung cancer, tuberculosis, bronchiectasis, pneumonia, acute bronchitis, cryptogenic haemoptysis or other causes. Epidemiology will be analysed related to the severity of the symptom (mild haemoptysis: drops of blood or bloody sputum; moderate haemoptysis: <500 ml/24 h, severe haemoptysis: 1-2 cups, as defined by Hirshberg et al. CHEST 1997).

SECONDARY OUTCOMES:
Sensitivity and specificity of chest X-ray, chest CT scan and bronchoscopy alone and in combination in the diagnosis of different causes of haemoptysis. | 18 months
  Sensitivity, specificity, positive and negative predictive values of of chest X-ray, computed tomography (CT) scan and bronchoscopy executed alone versus the combination of the exams in the diagnosis of different causes of haemoptysis (lung cancer, tuberculosis, bronchiectasis, pneumonia, acute bronchitis, cryptogenic haemoptysis and other causes).
Percentage and severity of recurrence of haemoptysis in the follow-up period. | 18 months
  Every patient will be followed with scheduled visits and phone calls for 18 months since the first episode of haemoptysis. The percentage of patient with recurrence of haemoptysis, the severity of recurrence, will be measured and analysed by descriptive statistics.
Sensitivity and specificity of bronchoscopy in localizing the bleeding side and lobe in relation to the timing of the haemoptysis. | 18 months
  Accuracy of bronchoscopy in localizing the side and the lobe source of the bleeding in relation to the timing of haemoptysis. The bronchoscopic findings will be analysed in relation to the timing of the bleeding (within 24 hours, between 24 and 48, 49 and 96 or over 96 hours after the occurrence of the symptom).
Patient survival in the follow-up period. | 18 months
  Every patient will be followed with scheduled visits and phone calls for 18 months since the first episode of haemoptysis. Patient survival will be measured and analysed by descriptive statistics.

OTHER OUTCOMES:
Prevalence of chronic obstructive pulmonary disease (COPD) in patients with haemoptysis by using spirometry with the threshold of FEV1/FVC <70 | 1 month or at clinical stability
  Prevalence of chronic obstructive pulmonary disease (COPD) in patients with haemoptysis will be assessed performing spirometry as described by European Respiratory Society Guidelines (European Respiratory Journal, 2005). COPD will be diagnosed in patient with a compatible clinical history (smoking history and frequent exacerbations) and the presence of a ventilatory obstructive defect as defined by a ratio of the forced expiratory volume in the first second and forced vital capacity (FEV1/FVC) <70.
Distribution of main causes of haemoptysis in the subgroup of patients undergoing medical therapies that increase the risk of bleeding. | 18 months
  To define the prevalence of diseases in patients presenting with haemoptysis in relation to the use of drugs such as antiaggregants or anticoagulants.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Mondoni, MD, Principal Investigator — Respiratory Unit, San Paolo Hospital, Dipartimento Scienze della Salute, Università degli Studi di Milano, Milan, Italy.; Paolo Carlucci, MD, Study Chair — Respiratory Unit, San Paolo Hospital, Dipartimento Scienze della Salute, Università degli Studi di Milano, Milan, Italy.; Stefano Centanni, MD, PhD, Study Director — Respiratory Unit, San Paolo Hospital, Dipartimento Scienze della Salute, Università degli Studi di Milano, Milan, Italy.
Locations (6):
- Italy (6):
  - Pneumologia, Azienda Ospedaliero Universitaria, Ancona
  - USC Pneumologia, Azienda Ospedaliera della Provincia di Lodi, Lodi
  - U.O. di Pnuemologia, Azienda Ospedaliera, Carlo Poma, Mantova
  - Respiratory Unit, San Paolo Hospital, Dipartimento Scienze della Salute, Università degli Studi di Milano., Milan
  - A.O.U. Maggiore della Carità - S.C.D.O. Pneumologia, Novara
  - Clinica Pneumotisiologica, AOU Sassari, Sassari

REFERENCES:
- [Derived] Mondoni M, Carlucci P, Cipolla G, Pagani M, Tursi F, Fois A, Pirina P, Canu S, Gasparini S, Bonifazi M, Marani S, Comel A, Saderi L, De Pascalis S, Alfano F, Centanni S, Sotgiu G. Long-term prognostic outcomes in patients with haemoptysis. Respir Res. 2021 Aug 4;22(1):219. doi: 10.1186/s12931-021-01809-6. PMID 34348724
- [Derived] Mondoni M, Carlucci P, Cipolla G, Fois A, Gasparini S, Marani S, Centanni S, Sotgiu G. Bronchoscopy to assess patients with hemoptysis: which is the optimal timing? BMC Pulm Med. 2019 Feb 11;19(1):36. doi: 10.1186/s12890-019-0795-9. PMID 30744616
- [Derived] Mondoni M, Carlucci P, Job S, Parazzini EM, Cipolla G, Pagani M, Tursi F, Negri L, Fois A, Canu S, Arcadu A, Pirina P, Bonifazi M, Gasparini S, Marani S, Comel AC, Ravenna F, Dore S, Alfano F, Sferrazza Papa GF, Di Marco F, Centanni S, Sotgiu G. Observational, multicentre study on the epidemiology of haemoptysis. Eur Respir J. 2018 Jan 4;51(1):1701813. doi: 10.1183/13993003.01813-2017. Print 2018 Jan. No abstract available. PMID 29301924